CLINICAL TRIAL: NCT06377930
Title: A Phase 2A, Multicenter, Open-label Study Evaluating the Safety and Efficacy of RAP-219 in Adult Participants With Refractory Focal Epilepsy
Brief Title: Study Evaluating the Safety and Efficacy of RAP-219 in Adult Participants With Refractory Focal Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rapport Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAP-219-FOS-201
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Focal Onset Seizures
Keywords: Epilepsy; RNS; long episode; FOS; Refractory focal epilepsy
MeSH Terms: conditions — Seizures; Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAP-219 (Experimental): Participants will receive 0.75 mg RAP-219 daily for 5 days followed by 1.25 mg RAP-219 daily for the remainder of the 8-week treatment period.
  Interventions: Drug: RAP-219

INTERVENTIONS:
Drug: RAP-219 — RAP-219 oral tablet

SUMMARY:
This is a clinical research study for an investigational drug called RAP-219 in patients with Refractory Focal Epilepsy. This study is being conducted to determine if RAP-219 works and is safe in patients with Refractory Focal Epilepsy.

DETAILED DESCRIPTION:
This is a Phase 2A, proof-of-concept, multi-center, open-label study designed to evaluate the efficacy, safety, tolerability, and PK/PD relationship of RAP-219 in adult participants with refractory focal epilepsy. The activity of RAP-219 will be assessed in approximately 30 participants treated with the RNS® system.

ELIGIBILITY:
Inclusion Criteria:

* Medically refractory focal epilepsy with an implanted responsive neurostimulator device placed correctly in a seizure onset zone that meet several device-related criteria and demonstrated history of compliance with interrogation of the RNS device and upload of data
* If currently treated with antiseizure medications, up to a maximum of 4 concomitant mediations are allowed
* At least 1 clinical seizure during the 8-week retrospective eligibility period
* Participants in otherwise good health as determined by the investigator
* Willing and able to adhere to all aspects of the protocol
* A demonstrated history of compliance with interrogation of the RNS device and upload of data before screening

Exclusion Criteria:

* Participants with generalized onset seizures in the past 10 years
* History of status epilepticus while on antiseizure medications within 2 years of screening
* Individuals of reproductive potential who do not agree to simultaneously use two effective birth-control methods
* Participants who have had epilepsy surgery within the last 12 months before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Change in long episode frequency during the treatment period compared to pre-treatment baseline: Responder proportion, Percent Change Percent change | Screening until 5 months after enrollment
  Change in long episode frequency per 28-day period during the treatment period compared to baseline

SECONDARY OUTCOMES:
Change in focal clinical seizure frequency during the treatment period compared to pre-treatment baseline: Percent Change, Responder proportion | Screening until 5 months after enrollment
  Change in focal clinical seizure frequency per 28-day period during the treatment period compared to baseline
Change in frequency of estimated electrographic seizures based on RNS® system data during the treatment period compared to pre-treatment baseline | Screening until 5 months after enrollment
  Change in the frequency per 28-day period of estimated electrographic seizures based on RNS data during the treatment period compared to baseline
Change in RNS® system long episode-free days during the treatment period compared to pre-treatment baseline: Count, Longest continuous interval, Time until pre-treatment count | Screening until 5 months after enrollment
  Change in long episode-free days during the treatment period compared to pre-treatment baseline
Change in focal clinical seizure-free days during the treatment period compared to pre-treatment baseline: Count, Longest continuous interval, Time until pre-treatment count | Screening until 5 months after enrollment
  Change in focal clinical seizure-free days during the treatment period compared to pre-treatment baseline
Change in RNS® system electrographic biomarkers other than long episodes during the treatment period compared to pre-treatment baseline | Dosing until 5 months after dosing
  Change in RNS® system electrographic biomarkers other than long episodes during the treatment period compared to pre-treatment baseline
Change in the Seizure Severity Response Questionnaire (SSRQ) during the treatment period compared to pre-treatment baseline | Screening until 5 months after enrollment
  Measurement of seizure severity by participant rating scale of the Seizure Severity Scale. Seizure severity will be assessed by asking participants to respond to 4 questions using a 0-10 numerical rating scale and circling the number that best describes how their seizures have impacted them since their last study visit. Higher scores = higher impact.
Count and proportion of responders on the clinical global impression of change (CGIC) scale during the treatment period compared to pre-treatment baseline | Screening until 5 months after enrollment
  Change in overall clinical status as measured by Clinical Global Impression of Change scores rated by investigator and participant. Both the participant (PGIC) and the clinician (CGIC) will rate their global impression of changes in the participant's condition throughout the study. The CGI scale measures the change in the participant's clinical status from a specific point in time, i.e., the Baseline Period and is rated on a 7-point Likert scale ranging from a score of 1 for very much improved to 7 for very much worse. Higher scores = worse outcome.
Plasma concentrations of RAP-219 | Dosing until 5 months after dosing
  Analysis of plasma concentrations of RAP-219
Incidence of treatment-emergent adverse events (TEAEs) | Dosing until 5 months after enrollment
  Analysis of AEs during the treatment and pre-treatment baseline periods
Clinically meaningful changes, if any, from baseline in vital signs, electrocardiograms (ECGs), complete blood counts, serum chemistries, or liver function tests after treatment with RAP-219 | Screening until 5 months after enrollment
  Analysis of vital signs, ECGs, CBC, serum chemistries and liver function tests during the treatment and pre-treatment baseline periods
Incidence of participants expressing suicidal ideation assessed with the Columbia-Suicide Severity Rating Scale (C-SSRS) | Screening until 5 months after enrollment
  Analysis of C-SSRS entries during the treatment and pre-treatment baseline periods
Cognitive function as measured using the Cogstate Digital Battery | Screening until 5 months after enrollment
  Analysis of the Cogstate Digital Battery during the treatment and pre-treatment baseline periods

CONTACTS AND LOCATIONS:
Overall Officials: Jaqueline A French, MD, Principal Investigator — NYU Langone Comprehensive Epilepsy Center
Locations (12):
- United States (12):
  - Yale University, New Haven, Connecticut
  - Consultants in Epilepsy and Neurology, PLLC, Boise, Idaho
  - IU Health Neuroscience Center, Goodman Hall, Indianapolis, Indiana
  - The University of Kansas Medical Center Epilepsy Clinic, Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Comprehensive Epilepsy Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania - Department of Neurology, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center, Houston, Houston, Texas